CLINICAL TRIAL: NCT01888510
Title: Comparison of Conventional Free Breathing CT, 4D CT, and Integrated Active Breath Hold CT Image Acquisition for Lung Cancer
Brief Title: CT in Diagnosing Patients With Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-15032; NCI-2013-01163 (Registry Identifier: NCI)
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (imaging studies) (Experimental): Patients undergo conventional free breathing CT, 4D CT, ABC CT, ABC CBCT, and free breathing CBCT before undergoing radiation therapy.
  Interventions: Procedure: computed tomography; Procedure: 4-dimensional computed tomography; Procedure: cone-beam computed tomography

INTERVENTIONS:
Procedure: computed tomography — Undergo conventional free breathing CT
  Other Names: tomography, computed
Procedure: 4-dimensional computed tomography — Undergo 4D CT
  Other Names: 4D-CT
Procedure: computed tomography — Undergo ABC CT
  Other Names: tomography, computed
Procedure: cone-beam computed tomography — Undergo ABC CBCT
Procedure: cone-beam computed tomography — Undergo free breathing CBCT

SUMMARY:
This clinical trial studies computed tomography (CT) in diagnosing patients with lung cancer. Diagnostic procedures, such as CT, may help find and diagnose lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct a prospective clinical imaging study to quantify the amount of inter- and intra-physician contouring variability on four dimensional (4D) CT, active breathing control (ABC) CT, free breathing CT, and free breathing and ABC cone beam (CB)CT.

II. Quantify the magnitude and distribution of target and organ at risk volume variations between the different imaging modalities.

III. Determine dosimetric changes related to contouring variations for tumor and normal tissue.

OUTLINE:

Patients undergo conventional free breathing CT, 4D CT, ABC CT, ABC CBCT, and free breathing CBCT before undergoing radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease on CT scan
* Patients with lung cancer visible on CT who are scheduled to receive external beam radiation treatment will be eligible for this study
* Patients must be able to perform ABC procedures

Exclusion Criteria:

* Patients requiring continuous supplemental oxygen due to the requirement of spirometry during all imaging studies
* No vulnerable populations will be enrolled (prisoners, children, pregnant females or institutionalized individuals)
* Women of childbearing potential will undergo a pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Amount of inter- and intra-physician contouring variability on 4D CT, ABC CT, free breathing CT, and free breathing and ABC CBCT | up to 1 week
  A two sided t-test with 5% level of significance will be used.

SECONDARY OUTCOMES:
Magnitude and distribution of target and organ at risk volume variations between the different imaging modalities | up to 1 week
  A two sided t-test with 5% level of significance will be used.
Dosimetric changes related to contouring variations for tumor and normal tissue | up to 1 week
  A two sided t-test with 5% level of significance will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Weiss, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States